CLINICAL TRIAL: NCT01761981
Title: Institutional Registry of Haemorrhagic Hereditary Telangiectasia
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MARCELO MARTIN SERRA, Marcelo Martin Serra, Hospital Italiano de Buenos Aires
Other Study IDs: 1900
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Haemorrhagic Hereditary Telangiectasia
Keywords: Haemorrhagic Hereditary Telangiectasia; Rendu Osler Weber Syndrome; Osler Weber Rendu Syndrome; HHT
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The purpose of this study is to create an institutional and population-based registry of Haemorrhagic Hereditary Telangiectasia with a prospective survey based on epidemiological data, risk factors, diagnosis, prognosis, treatment, monitoring and survival.

This study will also describe the occurrence of Haemorrhagic Hereditary Telangiectasia in the population of HIBA in the Central Hospital, as well as the characteristics of clinical presentation and evolution.

DETAILED DESCRIPTION:
Haemorrhagic Hereditary Telangiectasia is a uncommon autosomic hereditary disorder caracterizad for recurrent epistaxis,cutaneomucous telangiectasias and arteriovenous malformations in diferent organs; brain, lung, liver and gastrointestinal are more often afected . Afect one in 5000-8000 individual in worldwide. HHT may produce important morbidity like brain absces, stroke, hemoptisis and cronic ferropenic anemia.

Molecular mechanism of this disorder are complex and still no fully dilucidated. The genes mutated in HHT encode endothelial cell-expressed proteins that mediate signalling by the transforming growth factor (TGF)b superfamily. Endoglin (HHT type I) and ACVRL-1 (HHT type 2) mutations are responsible in more than 80% of the individuals. Mutation of SMAD 4 protein (MADH4)cause HHT in association with juvenile polyposis. HHT may associated with primary pulmonary hypertension en more rare cases.

There are not HHT registry in Argentina and Latinamerican population. This registry may gader valious information in order to generate a better diagnosis and treatment of our population and others.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HHT defined.
2. Followed in Unidad HHT of Hospital Italiano de Buenos Aires.

Exclusion Criteria:

1. Denied to participated in the registry or inform consent process.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Haemorrhagic Hereditary Telangiectasia
Sampling Method: Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
morbidity | 1 year
  Control visit every three month

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo M Serra, MD, Principal Investigator — HHT Center of Excelence Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serra MM, Besada CH, Cabana Cal A, Saenz A, Stefani CV, Bauso D, Golimstok AB, Bandi JC, Giunta DH, Elizondo CM. Central nervous system manganese induced lesions and clinical consequences in patients with hereditary hemorrhagic telangiectasia. Orphanet J Rare Dis. 2017 May 18;12(1):92. doi: 10.1186/s13023-017-0632-2. PMID 28521822